CLINICAL TRIAL: NCT06603038
Title: Perceived Wellbeing and Focus with Daily Greens Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gainful (Industry)
Responsible Party: Principal Investigator, Sarah Oliver, Manager, CRM and Retention, Gainful
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Gainful
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Well-Being, Psychological
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Supplementation with Daily Performance Greens daily for 28 days
  Interventions: Dietary Supplement: Gainful Daily Performance Greens
- Control (No Intervention): Control group, no supplementation

INTERVENTIONS:
Dietary Supplement: Gainful Daily Performance Greens — Daily supplementation for 28 days
  Arms: Intervention

SUMMARY:
This study aims to investigate whether daily consumption of Gainful Daily Performance Greens for four weeks contributes to improved scores of wellbeing and focus in healthy adults, as compared to a control group of non-supplement takers. The research question will be addressed by evaluating participants' responses using the World Health Organization's WHO-5 Wellbeing Index and the Mindful Attention Awareness Scale.

DETAILED DESCRIPTION:
Purpose: The primary objective of this study is to assess the potential benefits of Gainful Daily Performance Greens on wellbeing and focus in healthy adults. The formulation of this supplement includes ingredients believed to support mental clarity and overall wellbeing. Understanding the impact of this product on subjective measures of wellbeing and focus will provide valuable insights into its potential benefits for a broader population.

Hypotheses: H0 (null hypothesis): There is no significant difference in wellbeing and focus scores between baseline and after four weeks of daily Gainful Daily Performance Greens consumption in healthy adults. H1 (alternate hypothesis): Daily consumption of Gainful Daily Performance Greens for four weeks results in improved scores of wellbeing and focus as measured by the WHO-5 Wellbeing Index and Mindful Attention Awareness Scale compared to baseline in healthy adults.

Goals and Objectives: The primary goal is to examine the potential positive effects of Gainful Daily Performance Greens on wellbeing and focus. Specific objectives include comparing pre- and post-supplementation scores using validated measures, identifying any changes in subjective experiences related to mental clarity and wellbeing, and exploring potential factors influencing individual responses.

Significance of Study: Understanding the impact of Gainful Daily Performance Greens on wellbeing and focus addresses the growing interest in functional foods and dietary supplements. If the study demonstrates positive effects, it may provide evidence for the inclusion of such supplements in promoting overall mental health and wellbeing in healthy adults.

Contribution to Field: This study contributes to the emerging field of nutritional interventions for overall wellbeing. By using established scales to measure wellbeing and focus, the research aims to provide valuable insights into the potential benefits of Gainful Daily Performance Greens, informing future research and dietary recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Not currently taking cognitive-enhancing supplements or medications
* Provide informed consent
* Have the ability to comply with the study protocol

Exclusion Criteria:

* Known allergy to the ingredients of Daily Performance Greens

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2024-04-26 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Perceived Wellbeing | 28 days
  Measured using WHO-5 Wellbeing Index Scale (0-5, where 5 is better outcome)
Mindfulness | 28 days
  Measured using Mindful Attention Awareness Scale (1-6, where 6 is better outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Gainful, New York, New York, United States